CLINICAL TRIAL: NCT05936151
Title: A Phase 2b, Double-Blind Study to Investigate the Effect of Retatrutide on Renal Function in Participants With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes
Brief Title: A Study of Retatrutide (LY3437943) on Renal Function in Participants With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18725; J1I-MC-GZBU (Other: Eli Lilly and Company); 2023-504583-42-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Overweight or Obesity; CKD; Type 2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2b
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Retatrutide (Experimental): Participants will receive multiple doses of retatrutide subcutaneously (SC)
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive LY3437943
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the effect of retatrutide on renal function in participants with overweight or obesity and chronic kidney disease (CKD), with or without Type 2 Diabetes (T2D). The study will last around 31 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥27 kilogram/square meter (kg/m²)
* Have either

  * no T2D with an HbA1c < 6.5% or
  * have T2D with an HbA1c ≤ 9.5% and treated with diet and exercise only or with stable doses of up to 3 oral antihyperglycemic medications, with or without basal insulin for at least 90 days before screening.
* Have been diagnosed with chronic kidney disease (CKD).

Exclusion Criteria:

* Have a self-reported change in body weight >5 kilogram (kg) (11 pounds) within 90 days before screening.
* Have used in 90 days before the screening any of the following antihyperglycemic class: Dipeptidyl Peptidase IV (DPP4) inhibitors, amylin analogs, glucagon-like peptide-RA (GLP-RA), gastric inhibitory polypeptide (GIP)/GIP-1 RA, and short acting or rapid acting insulins or U500 Insulin
* Have a prior or planned surgical treatment for obesity
* Have Type 1 Diabetes (T1D)
* Have acute or chronic hepatitis
* Have a history of malignant disease within 5 years before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glomerular Filtration Rate (mGFR) | Baseline, Week 24
  The GFR in milliliter/minute per1.73 square meter (mL/min/1.73 m²) using iohexol clearance (mGFR-measured glomerular filtration rate)

SECONDARY OUTCOMES:
Change from Baseline in Urine Albumin-to-Creatinine Ratio (UACR) | Baseline, Week 24
Change from Baseline in Creatinine-Corrected Fractional Urinary Sodium Excretion (FENa) | Baseline, Week 24
Change from Baseline in Filtration Fraction Estimated from Measured Glomerular Filtration Rate (mGFR) | Baseline, Week 24
Change from Baseline in Renal Mean Arterial Flow as Assessed by Magnetic Resonance Imaging (MRI), Corrected by Hematocrit | Baseline, Week 24
Change from Baseline in in Mean Arterial Flow (MAF) | Baseline, Week 24
Change from Baseline in Renal Artery Resistive Index (RARI) | Baseline, Week 24
Change from Baseline in Renal Blood Flow Velocity Peak Systolic Velocity (PSV) and End-diastolic Velocity (ESV) | Baseline, Week 24
Change from Baseline in Global Renal Perfusion (MRI) | Baseline, Week 24
Change from Baseline in Total Renal Parenchyma Volume (MRI) | Baseline, Week 24
Change from Baseline in Renal Cortex Volume (MRI) | Baseline, Week 24
Change from Baseline in Renal Cortex T1 (ms) (MRI) | Baseline, Week 24
Change from Baseline in Medulla T1 (ms) (MRI) | Baseline, Week 24
Change from Baseline in Renal Cortex R2 (BOLD MRI) | Baseline, Week 24
Change from Baseline in Medulla R2 | Baseline, Week 24
Change from Baseline in Body Weight | Baseline, Week 24
Change from Baseline in 24-hr Urinary Albumin Excretion (UAE) | Baseline, Week 24
Change from Baseline in Change in 24-hour (hr) Urinary Electrolytes (milligrams/24hr (mg/24h)) | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (42):
- United States (19):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - Care Access - 801 South Power Road, Mesa, Mesa, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Medical Advancement Centers of Arizona, Tempe, Arizona
  - Hope Clinical Research, Inc., Canoga Park, California
  - Catalina Research Institute, LLC, Montclair, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Teradan Clinical Trials, LLC, Brandon, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Prime Health and Wellness/SKYCRNG, Fayette, Mississippi
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Victorium Clinical Research - Houston, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Tranquility Research, Webster, Texas
- Canada (9):
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Circulate Cardiac & Vascular Centre, Burlington, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Fadia El Boreky Medicine, Waterloo, Ontario
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - Diex Recherche Joliette, Joliette, Quebec
  - 9109-0126 Quebec Inc., Montreal, Quebec
- Italy (4):
  - Centro Cardiologico Monzino, Milan, Milano
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Ospedale San Raffaele, Milan
- Spain (3):
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Doctor Peset, Valencia, Valenciana, Comunitat
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - FutureMeds Teesside - Middlefield Centre, Stockton-on-Tees, Durham County
  - Royal London Hospital, London, England
  - Futuremeds-Newcastle, Newcastle, England
  - Vascular Research Team, Salford, Greater Manchester
  - North Middlesex Hospital, London, London, City of
  - City Hospital, Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) on Renal Function in Participants With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes — https://trials.lilly.com/en-US/trial/410437.